CLINICAL TRIAL: NCT01008930
Title: Feasibility Study for Imaging of Peripheral Tumors With a High-Resolution PET Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2009-0478; NCI-2011-02894 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Solid Tumors; Cancer
Keywords: Peripheral Tumors; Arm; Leg; Head; Neck; HR PET Imaging System; High-Resolution PET; PET/CT; PEMFlex Solo II; positron emission tomography/computed tomography (PET/CT)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEM Scan (Experimental): HR PEM images (High Resolution PEMFlex Solo II scan images)
  Interventions: Procedure: HR PEM Scan

INTERVENTIONS:
Procedure: HR PEM Scan — PEMFlex Solo II, a high-resolution camera for PET scan imaging, on an area of body that has, or is suspected to have cancer following routine, standard, positron emission tomography/computed tomography (PET/CT) scan
  Other Names: HR PET/CT Scan; PET/CT Imaging; PET; CT; Computed Tomography

SUMMARY:
The goal of this clinical research study is to learn if using the PEMFlex Solo II, a high-resolution camera for PET scan imaging, on an area of the body that has, or is suspected to have cancer will give researchers the same or better information about the disease compared to the images taken with a routine PET/CT.

Researchers will compare the images taken using the PEMFlex Solo II to the images taken during your scheduled routine PET/CT scan, as well as any additional routine CT scan(s), magnetic resonance imaging (MRI) scan(s), and/or ultrasound image(s) you may have had within the last 30 days or may have in the next 30 days.

DETAILED DESCRIPTION:
If you agree to take part in this study, right after your already-scheduled routine PET/CT scan is complete, a study staff member will take you to a separate imaging room located in the same clinic area where your routine PET/CT scan was just performed.

You will then sit in a chair as a study staff member positions the PEMFlex Solo II on either side of the area being checked for cancer. It will take about 20 minutes to set up the PEMFlex Solo II and take the PET scan images.

Length of Study:

After the PET scan images have been taken using the PEMFlex Solo II, your participation in this study will be over.

This is an investigational study. The PEMFlex Solo II is commercially available and designed for PET scan imaging of the breast. The use of the PEMFlex Solo II for imaging other parts of the body is investigational.

Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent.
2. Known or suspected primary or metastatic lesion of the extremities, head or neck as determined by biopsy, physical examination or noninvasive imaging studies including plain films, CT, MR, ultrasound or nuclear medicine imaging.
3. Scheduled for routine clinical imaging at the ACB PET/CT facility.
4. Participant must be at least 18 years of age.

Exclusion Criteria:

1. Uncontrolled blood glucose levels (>200 mg/dl).
2. Patient is unable to comprehend the requirements of the study.
3. Patient is unable to undergo scanning of the known or suspected lesion with the high-resolution PEM (PET) scanner (due to body habitus, inability to comply with positioning requirements, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of peripheral tumor lesions identified in standard PET/CT imaging also identifiable in PEM images. | 20 minutes for imaging using PEMFlex Solo II
  Study considered a success if 70% of lesions identified using standard images are also identifiable in the PEM image.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rohren, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org